CLINICAL TRIAL: NCT04182997
Title: Subjective Intraoperative Use of Epidural Steroid Administration Following Discectomy for Herniated Lumbar Discs Is There a Role? - A Randomized Control Trial
Brief Title: Subjective Intraoperative Use of Epidural Steroid Administration Following Discectomy
Acronym: Intra-Op
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Don Moore, MD, Assistant Professor, Orthopedic Surgery, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014147
Record Dates: First submitted 2019-11-25; First posted 2019-12-02 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Dexamethasone; Calcium Dobesilate; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to either the treatment group or the placebo group. At the end of surgery patients in the treatment group will have the surgical site lavaged with dexamethasone while patients in the placebo group will have the surgical site lavaged by sterile saline.
Who Masked: Participant
Masking Description: The patient will be blinded to which arm they were assigned. This will be accomplished by the research coordinator determining the randomization status and passing this information along to a surgical nursing staff. The nurse will the procure either the placebo or treatment drug and give it to the treating physician and announce which treatment drug the patient is receiving.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo Group (Placebo Comparator): Patients in this group will be given the placebo (sterile saline).
  Interventions: Drug: saline 0.9%
- Dexamethasone Group (Active Comparator): Patients in this group will be given the study drug (dexamethasone).
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Patients included in the treatment group will have their surgical site lavaged with dexamethasone at the end of their surgery.
  Other Names: Decadron
  Arms: Dexamethasone Group
Drug: saline 0.9% — Patients included in the placebo group will have their surgical site lavaged with sterile saline at the end of their surgery.
  Other Names: sterile saline
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to determine a grading system for inflammation in lumbar disc herniation and which groups, if any, benefit most from the administration of an intra-operative epidural steroid.

DETAILED DESCRIPTION:
Intraoperative epidural administration of steroids following discectomy for herniated lumbar disc has been the topic of multiple studies in the literature. The results have been mixed, with the majority of the studies finding some benefit, but outcomes have varied drastically amongst the many studies. The aim of this study is to develop a grading scale for intraoperative assessment of nerve root inflammation to determine if this subjective assessment is an adequate indicator for response to epidural steroids following discectomy. Patients will be allocated randomly preoperatively to the intervention group versus control group. Pictures of the spinal cord and associated nerve root will be captured intraoperatively. These pictures will be scrutinized postoperatively and an inflammation grade will be assigned. The investigators will then identify if nerve roots with a higher-grade of inflammation respond differently to epidural steroid administration when compared to lesser-grades of inflammation. This will be measured with the a variety of outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to the University of Missouri hospital system - including the University of Missouri Hospital and Missouri Orthopaedic Institute - with a clinical assessment indicative of a lumbar disc herniation
* Failed conservative treatment - rest, anti-inflammatory medications, physical therapy
* Radiculopathy present - positive tension signs or sensory/motor neurologic deficits present
* Recent MRI confirming single-level lumbar disc herniation corresponding to clinical evaluation

Exclusion Criteria:

* Concomitant spinal stenosis, segmental instability, or spondylolisthesis
* Previous surgery at the affected level or recurrent herniation
* Underlying disease that may affect response to steroids - immunocompromise, use of chronic steroids or immunosuppression
* Pregnancy - qualitative human chorionic gonadotropin (hCG) testing will be performed prior to enrollment
* Diagnosis of or symptoms concerning for cauda equina syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-11-21 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Post Operative Pain Scores | Until final follow up (up to 8 weeks)
  Comparing post operative pain scores between treatment and placebo group. Using Visual Analogue Scale (VAS) pain score with scale 0 to 10 with 0 being no pain and 10 being the worst pain of your life.
Post Operative Oswestry Disability Index | Until final follow up (up to 8 weeks
  Comparing post operative disability scores between treatment and placebo group. Using Oswestry Disability Index (ODI) to measure a patient's permanent functional disability and low back functional outcome tools.

SECONDARY OUTCOMES:
Length of stay | Until final follow up (up to 8 weeks)
  Determining how long patient is in hospital
Post Operative Opioid Usage | Until final follow up (up to 8 weeks)
  comparing opioid usage post operatively
Post Operative Complications | Until final follow up (up to 8 weeks)
  comparing rate of post-op infections

CONTACTS AND LOCATIONS:
Overall Officials: Don Kim Moore, MD, Principal Investigator — Missouri Orthopaedic Institute
Locations (1):
- Missouri Orthopaedic Institute, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akinduro OO, Miller BA, Haussen DC, Pradilla G, Ahmad FU. Complications of intraoperative epidural steroid use in lumbar discectomy: a systematic review and meta-analysis. Neurosurg Focus. 2015 Oct;39(4):E12. doi: 10.3171/2015.7.FOCUS15269. PMID 26424336
- [Background] Aljabi Y, El-Shawarby A, Cawley DT, Aherne T. Effect of epidural methylprednisolone on post-operative pain and length of hospital stay in patients undergoing lumbar microdiscectomy. Surgeon. 2015 Oct;13(5):245-9. doi: 10.1016/j.surge.2014.03.012. Epub 2014 Jun 7. PMID 24916651
- [Background] Arirachakaran A, Siripaiboonkij M, Pairuchvej S, Setrkraising K, Pruttikul P, Piyasakulkaew C, Kongtharvonskul J. Comparative outcomes of epidural steroids versus placebo after lumbar discectomy in lumbar disc herniation: a systematic review and meta-analysis of randomized controlled trials. Eur J Orthop Surg Traumatol. 2018 Dec;28(8):1589-1599. doi: 10.1007/s00590-018-2229-4. Epub 2018 May 29. PMID 29845327
- [Background] Debi R, Halperin N, Mirovsky Y. Local application of steroids following lumbar discectomy. J Spinal Disord Tech. 2002 Aug;15(4):273-6. doi: 10.1097/00024720-200208000-00002. PMID 12177541
- [Background] Diaz RJ, Myles ST, Hurlbert RJ. Evaluation of epidural analgesic paste components in lumbar decompressive surgery: a randomized double-blind controlled trial. Neurosurgery. 2012 Feb;70(2):414-23; discussion 423-4. doi: 10.1227/NEU.0b013e3182315f05. PMID 21841518
- [Background] Jamjoom BA, Jamjoom AB. Efficacy of intraoperative epidural steroids in lumbar discectomy: a systematic review. BMC Musculoskelet Disord. 2014 May 5;15:146. doi: 10.1186/1471-2474-15-146. PMID 24885519
- [Background] Jirarattanaphochai K, Jung S, Thienthong S, Krisanaprakornkit W, Sumananont C. Peridural methylprednisolone and wound infiltration with bupivacaine for postoperative pain control after posterior lumbar spine surgery: a randomized double-blinded placebo-controlled trial. Spine (Phila Pa 1976). 2007 Mar 15;32(6):609-16; discussion 617. doi: 10.1097/01.brs.0000257541.91728.a1. PMID 17413463
- [Background] Karst M, Kegel T, Lukas A, Ludemann W, Hussein S, Piepenbrock S. Effect of celecoxib and dexamethasone on postoperative pain after lumbar disc surgery. Neurosurgery. 2003 Aug;53(2):331-6; discussion 336-7. doi: 10.1227/01.neu.0000073530.81765.6b. PMID 12925248
- [Background] Kennedy DJ, Zheng PZ, Smuck M, McCormick ZL, Huynh L, Schneider BJ. A minimum of 5-year follow-up after lumbar transforaminal epidural steroid injections in patients with lumbar radicular pain due to intervertebral disc herniation. Spine J. 2018 Jan;18(1):29-35. doi: 10.1016/j.spinee.2017.08.264. Epub 2017 Sep 28. PMID 28962912
- [Background] Keorochana G, Pairuchvej S, Setrkraising K, Arirachakaran A, Kongtharvonskul J. Comparative Outcomes of Perioperative Epidural Steroids After Percutaneous Endoscopic Lumbar Discectomy for Lumbar Disc Herniation: A Randomized Placebo-Controlled Trial. World Neurosurg. 2018 Nov;119:e244-e249. doi: 10.1016/j.wneu.2018.07.122. Epub 2018 Jul 27. PMID 30059778
- [Background] Mirzai H, Tekin I, Alincak H. Perioperative use of corticosteroid and bupivacaine combination in lumbar disc surgery: a randomized controlled trial. Spine (Phila Pa 1976). 2002 Feb 15;27(4):343-6. doi: 10.1097/00007632-200202150-00003. PMID 11840097
- [Background] Rasmussen S, Krum-Moller DS, Lauridsen LR, Jensen SE, Mandoe H, Gerlif C, Kehlet H. Epidural steroid following discectomy for herniated lumbar disc reduces neurological impairment and enhances recovery: a randomized study with two-year follow-up. Spine (Phila Pa 1976). 2008 Sep 1;33(19):2028-33. doi: 10.1097/BRS.0b013e3181833903. PMID 18758356
- [Background] Shin SH, Hwang BW, Keum HJ, Lee SJ, Park SJ, Lee SH. Epidural Steroids After a Percutaneous Endoscopic Lumbar Discectomy. Spine (Phila Pa 1976). 2015 Aug 1;40(15):E859-65. doi: 10.1097/BRS.0000000000000990. PMID 25996534
- [Background] Wilson-Smith A, Chang N, Lu VM, Mobbs RJ, Fadhil M, Lloyd D, Kim S, Phan K. Epidural Steroids at Closure After Microdiscectomy/Laminectomy for Reduction of Postoperative Analgesia: Systematic Review and Meta-Analysis. World Neurosurg. 2018 Feb;110:e212-e221. doi: 10.1016/j.wneu.2017.10.133. Epub 2017 Nov 1. PMID 29102751